CLINICAL TRIAL: NCT04071132
Title: Using Adhesive Biosensor Patches to Characterize the Biochemical Phenotype in Individuals Diagnosed With PTSD
Brief Title: Using Adhesive Biosensor Patches to Characterize the Biochemical Phenotype in PTSD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nadav Goldental (Other)
Responsible Party: Sponsor-Investigator, Nadav Goldental, Principal investigator, The Chaim Sheba Medical Center
Organization: The Chaim Sheba Medical Center (Other)
Other Study IDs: 6381-19-SMC
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants diagnosed with PTSD
- Non-PTSD participants

SUMMARY:
A psychiatric diagnosis of post-traumatic stress disorder (PTSD) is currently based mainly on non-quantitative elements, such as interviews and subjective impressions. PTSD has physiological manifestations, some of which are likely reflected in the levels and ratios of certain stress-related proteins in the interstitial fluid and plasma. Discernable patterns of such stress-related proteins may constitute a biochemical phenotype characteristic of PTSD, which may serve as a biomarker and support diagnostic decisions, as well as personalized treatment plans.

The current study is a non-interventional observational study aimed at examining the possibility of basing a psychiatric diagnosis by measuring changes in the biochemical phenotype of participants with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis (excluding controls)
* Proper ability to give informed consent

Exclusion Criteria:

* Active psychotic or suicidal symptoms
* Active/terminal oncological condition
* Dialysis patients
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult (aged 18 and over) participants with and without PTSD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Changes in cortisol levels | 3 months
  Changes in cortisol levels as measured by the adhesive biosensor patches
Changes in c-reactive protein (CRP) | 3 months
  Changes in c-reactive protein (CRP) levels as measured by the adhesive biosensor patches
Changes in Interleukin 6 (IL-6) levels | 3 months
  Changes in Interleukin 6 (IL-6) levels as measured by the adhesive biosensor patches
Changes in N-terminal pro b-type Natriuretic Peptide (NT-proBNP) levels | 3 months
  Changes in N-terminal pro b-type Natriuretic Peptide (NT-proBNP) levels as measured by the adhesive biosensor patches
Changes in 8-Oxo-2'-deoxyguanosine (8-oxo-dg) levels | 3 months
  Changes in 8-Oxo-2'-deoxyguanosine (8-oxo-dg) levels as measured by the adhesive biosensor patches
Changes in volatile organic compounds (VOCs) levels | 3 months
  Changes in volatile organic compounds (VOCs) concentrations (hexanone, acetic acid, heptane, hexanal, 3-heptanone, hexanoic acid, heptanal and nonanal) as measured by the adhesive biosensor patches
Changes in glucose levels | 3 months
  Changes in glucose levels as measured by the adhesive biosensor patches
Correlations between biochemical changes and PTSD clinical symptoms | 3 months
  Correlations between biochemical changes and questionnaire data relating to PTSD clinical symptoms (CGI, CAPS, PHQ, PCL-5, PC-PTSD-5, LEC-5 and BARS).